CLINICAL TRIAL: NCT05629806
Title: Effect of Acarbose and Fixed Mixture of Pioglitazone and Metformin in Patients With Type 2 Diabetes Receiving Anti-diabetic Monotherapy
Brief Title: Effect of Acarbose and Mixture of Pioglitazone and Metformin in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KY20220314-02
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Type 2 Diabetes; Blood Glucose Fluctuation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone; Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin plus pioglitazone (Active Comparator)
  Interventions: Drug: Metformin plus pioglitazone; Drug: Acarbose
- Acarbose (Active Comparator)
  Interventions: Drug: Metformin plus pioglitazone; Drug: Acarbose

INTERVENTIONS:
Drug: Metformin plus pioglitazone — After the screening period, eligible subjects were admitted to two tablets of fixed mixture of metformin plus pioglitazone (15mg pioglitazone plus 500mg metformin) for 12 weeks. Then the subjects were titrated onto the alternative treatment of 50mg acarbose three times daily for 12 weeks. During this timeframe, all patients were instructed to monitor their blood glucose fluctuations with a FreeStyle Libre Pro Sensor (FGM system) before and after the study and the time point of drug replacement.
Drug: Acarbose — After the screening period, eligible subjects were admitted to 50mg acarbose three times daily for 12 weeks. Then the subjects were titrated onto the alternative treatment of two tablets of fixed mixture of metformin plus pioglitazone (15mg pioglitazone plus 500mg metformin) for 12 weeks. During this timeframe, all patients were instructed to monitor their blood glucose fluctuations with a FreeStyle Libre Pro Sensor (FGM system) before and after the study and the time point of drug replacement.

SUMMARY:
Monotherapy with DPP-IV inhibitors, SGLT-2 inhibitors or insulin secretagogues frequently failed to maintain blood glucose in patients with type 2 diabtes. It was critical to determine which was more suitable of acarbose versus metformin plus pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in this present study;
* Patients with type 2 diabetes receiving stable monotherapy of DPP-IV inhibitors, SGLT-2 inhibitors or insulin secretagogues for more than 3 months;
* Screening glycated hemoglobin (HbA1c) between 7.0% and 10.0%;
* Regular diet and exercise;
* Body mass index (BMI) ≥ 18.5 kg/m2

Exclusion Criteria:

* Intolerance of metformin, pioglitazone and acarbose;
* Severe liver disease or elevated transaminases (2.5-fold the upper limit);
* Renal dysfunction or elevated creatinine (1.3-fold the upper limit);
* Systemic steroids therapy or other medication influencing cholesterol metabolism in the past 3 months;
* Infection or stress state in the past 4 weeks;
* Pregnancy or lactation;
* Patients otherwise adjudged by the investigator to be inappropriate for inclusion into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose fluctuation | week 24
  change from baseline blood glucsoe fluctuation at end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, China

IPD SHARING:
Plan to Share IPD: No